CLINICAL TRIAL: NCT03981562
Title: Vitamin D Supplementation and Reduction of Severity and Frequency of Epistaxis in Hereditary Haemorrhagic Telangiectasia
Brief Title: Vitamin D and Hereditary Haemorrhagic Telangiectasia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Paul's Hospital, Canada (Other)
Responsible Party: Principal Investigator, Amin Javer, Director, St. Paul's Sinus Centre, St. Paul's Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H18-01337
Record Dates: First submitted 2019-05-24; First posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Hereditary Haemorrhagic Telangiectasia
Keywords: Epistaxis
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Epistaxis

STUDY DESIGN:
Intervention Model Description: Patients included in the study will be randomized. Block randomization will be utilized to ensure an equal number of experimental and control patients are in each arm. A closed envelope system will be used to randomize participants within each arm.
Who Masked: Participant, Investigator
Masking Description: The study is double blinded, the investigators and the patients throughout the data collection and data analysis period will not be aware of the vitamin D dosage given.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1000 IU Vitamin D (Experimental)
  Interventions: Drug: Vit D
- 4000 IU Vitamin D (Experimental)
  Interventions: Drug: Vit D
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Vit D — Patients will take an oral vitamin D supplement once a day for 6 months.
  Arms: 1000 IU Vitamin D; 4000 IU Vitamin D
Drug: Placebo Oral Tablet — Patients will take a placebo oral tablet once a day for 6 months.
  Arms: Placebo

SUMMARY:
The study aims to assess whether supplementing vitamin D in patients diagnosed with Hereditary Haemorrhagic Telangiectasia (HHT) will decrease the frequency and severity of nosebleeds these patients experience. It is hypothesized that the larger the dose of daily vitamin D given to the patients, the less frequent and less severe the nosebleeds will be.

DETAILED DESCRIPTION:
1. Purpose:

   The focus of the study is to determine if supplementing vitamin D in patients diagnosed with HHT will reduce the frequency and severity of epistaxis episodes.
2. Hypothesis:

   For patients diagnosed with HHT, daily vitamin D supplementation will reduce the frequency and severity of epistaxis. Additionally, there will be a greater reduction in epistaxis frequency and severity the larger the dose of daily vitamin D supplemented
3. Justification:

   Hereditary haemorrhagic telangiectasia (HHT) is a rare autosomal dominant inherited disorder of the fibrovascular tissue that causes malformation of capillaries (called "telangiectases") and/or larger blood vessels (called "arteriovenous malformations") throughout the body. The formation of these lesions ultimately result in patients experiencing increased tendency for bleeding. These lesions may present in varying locations systemically, however recurrent and severe epistaxis is the most common presentation of HHT.

   Various medical and surgical treatments exist for management of HHT patients which are aimed at decreasing the frequency and severity of epistaxis episodes. These therapies include: humidification, nasal lubrication, nasal hot saline irrigation, intranasal packing, oestrogen ointment, tranexamic acid, bevacizumab systemic/topically applied, use of propranolol to lower blood pressure, electrocautery and YAG laser. Although all these various options are available, there currently is no consensus toward an optimal solution. Treatment can become especially difficult due to progressive anaemia or when anticoagulant or anti-thrombotic therapy becomes necessary. Therefore, there is a need for establishment of a safe and effective therapy.

   It has been suggested that vitamin D plays a role in cardiovascular health. Vitamin D plays a key role in establishing the integrity of blood vessels as it has been shown to provide protection of the vascular wall as well has having minor anticoagulation effects. As well, observational retrospective studies have found an association between vitamin D levels and epistaxis bleeding time and severity in HHT patients, with higher serum vitamin D levels being associated with decrease epistaxis bleeding time and severity. Despite evidence of positive effect of vitamin D on HHT, currently no prospective study has been done.
4. Objectives:

   Primary Objective To determine if vitamin D supplementation with 1000 IU or 4000 IU will reduce the frequency and severity of epistaxis in HHT patients.

   Secondary Objective To determine the adequate dosage of vitamin D supplementation required to reduce frequency and severity of epistaxis in HHT patients.
5. Research Method

The proposed study is a prospective double-blinded, placebo controlled, randomized control trial.

All the St. Paul's Sinus Centre patients willing to participate in the study will be invited for screening. Currently, the clinic has ~60 patients with HHT; therefore the investigators hope to enrol ~20 patients in each of the three study arms.

Consenting patient will be randomized to ensure equal number of experimental and control patients are in each arm. A closed envelop system will be used to randomize participants within each arm. Patients diagnosed with HHT who are not taking vitamin D supplementation at the time of recruitment will be randomized into one of the following three groups:

1. 1000 IU/day vitamin D,
2. 4000 IU/day vitamin D, or
3. Placebo control Patients who are already taking vitamin D at the time of recruitment will be asked to stop taking the current dose of vitamin D and will be randomized into either the 1000 IU or 4000 IU arm of the study. Patients previously taking Vitamin D will not participate as placebo controls.

Upon enrolment in the study, demographic data will be obtained, including age, gender, and ethnicity. Patient's will also have baseline blood work drawn, standard of care, (full hematological profile, ferritin, aPTT, INR, serum vitamin D, IgE) and be asked to fill out a questionnaire to provide a baseline Epistaxis Severity Score (ESS). This questionnaire is routinely used to assess quality of life in HHT patients and includes six independent predictors of self-described epistaxis severity. Baseline nasal endoscopic scoring will also be performed by endoscopic imaging of the nasal cavity.

The patients will be instructed on dosing of vitamin D supplementation. Patients will continue daily supplementation for three months until the first follow up visit. At the first follow-up visit patients will again have blood work drawn, be asked to fill out the ESS questionnaire, and receive nasal endoscopic scoring.

The last follow-up visit will be at six months and a repeat of the same procedures/tests will be carried out.

6. Statistical Analysis:

The primary outcome of this study will be the Epistaxis Severity Score (ESS), which is obtained from patient questionnaires. The secondary outcome will be the Nasal Endoscopic Score. The difference in the ESS and endoscopic score before and after supplementation within and between groups will be analyzed using paired and unpaired students t-tests based on the variance results.

Descriptive statistics (mean, median, SD) will be used to describe demographic and hematological data collected.

ELIGIBILITY:
Inclusion Criteria:

* 19 years or older
* Definite diagnosis of HHT using the Curacao criteria;
* HHT patients already on Vitamin D supplementation (these patients will still be included since the study is examining mega-doses specifically)

Exclusion Criteria:

* Patients with sinonasal tumours;
* Patients with bleeding disorders;
* Patients with serum levels of 250 or more ng/ml of vitamin D before or during the study supplementation (considered to be toxic levels)
* Patients who are unable to speak English;
* Patients who live outside B.C.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-07-16 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Epistaxis Severity Score | Baseline, 3 months, and 6 months
  A questionnaire that will be given to the patients at each visit which is a major predictor of quality of life in HHT patients.
  The score includes six independent predictors of self-described epistaxis severity. The responses will then be weighted by respective coefficients and these added together to give a raw ESS, which will then be divided by the range of the raw score (2.71) and multiplied by 10 to give normalized ESS within the range of 0 to 10 (no epistaxis to severe epistaxis).

SECONDARY OUTCOMES:
Change in Modified Lund-Kennedy Score | Baseline, 3 months, and 6 months
  The score is an objective measure based on Endoscopic sinonasal mucosal inflammation. The score is determined from a range of 0-12 with higher numbers indicating worse inflammation. Endoscopy will determine the density and location of telangiectasias, vascular morphology or patterns, relative percentage of arteriovenous malformations (AVMs), degree of crusting, septal perforation and site.

CONTACTS AND LOCATIONS:
Locations (1):
- E.N.T Clinic, St. Paul's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available to other researchers.

REFERENCES:
- [Background] Govani FS, Shovlin CL. Hereditary haemorrhagic telangiectasia: a clinical and scientific review. Eur J Hum Genet. 2009 Jul;17(7):860-71. doi: 10.1038/ejhg.2009.35. Epub 2009 Apr 1. PMID 19337313
- [Background] Shovlin CL, Guttmacher AE, Buscarini E, Faughnan ME, Hyland RH, Westermann CJ, Kjeldsen AD, Plauchu H. Diagnostic criteria for hereditary hemorrhagic telangiectasia (Rendu-Osler-Weber syndrome). Am J Med Genet. 2000 Mar 6;91(1):66-7. doi: 10.1002/(sici)1096-8628(20000306)91:13.0.co;2-p. PMID 10751092
- [Background] Hoag JB, Terry P, Mitchell S, Reh D, Merlo CA. An epistaxis severity score for hereditary hemorrhagic telangiectasia. Laryngoscope. 2010 Apr;120(4):838-43. doi: 10.1002/lary.20818. PMID 20087969
- [Background] Chamali B, Finnamore H, Manning R, Laffan MA, Hickson M, Whelan K, Shovlin CL. Dietary supplement use and nosebleeds in hereditary haemorrhagic telangiectasia - an observational study. Intractable Rare Dis Res. 2016 May;5(2):109-13. doi: 10.5582/irdr.2016.01019. PMID 27195194
- [Background] Plauchu H, de Chadarevian JP, Bideau A, Robert JM. Age-related clinical profile of hereditary hemorrhagic telangiectasia in an epidemiologically recruited population. Am J Med Genet. 1989 Mar;32(3):291-7. doi: 10.1002/ajmg.1320320302. PMID 2729347
- [Background] Al Mheid I, Patel R, Murrow J, Morris A, Rahman A, Fike L, Kavtaradze N, Uphoff I, Hooper C, Tangpricha V, Alexander RW, Brigham K, Quyyumi AA. Vitamin D status is associated with arterial stiffness and vascular dysfunction in healthy humans. J Am Coll Cardiol. 2011 Jul 5;58(2):186-92. doi: 10.1016/j.jacc.2011.02.051. PMID 21718915
- [Background] Min B. Effects of vitamin d on blood pressure and endothelial function. Korean J Physiol Pharmacol. 2013 Oct;17(5):385-92. doi: 10.4196/kjpp.2013.17.5.385. Epub 2013 Oct 17. PMID 24227938
- [Background] Weber LM, McDonald J, Whitehead K. Vitamin D levels are associated with epistaxis severity and bleeding duration in hereditary hemorrhagic telangiectasia. Biomark Med. 2018 Apr;12(4):365-371. doi: 10.2217/bmm-2017-0229. Epub 2018 Mar 14. PMID 29537299
- [Background] Geisthoff UW, Nguyen HL, Roth A, Seyfert U. How to manage patients with hereditary haemorrhagic telangiectasia. Br J Haematol. 2015 Nov;171(4):443-52. doi: 10.1111/bjh.13606. Epub 2015 Jul 23. PMID 26205234
- [Background] McDonald J, Bayrak-Toydemir P, Pyeritz RE. Hereditary hemorrhagic telangiectasia: an overview of diagnosis, management, and pathogenesis. Genet Med. 2011 Jul;13(7):607-16. doi: 10.1097/GIM.0b013e3182136d32. PMID 21546842
- [Background] Reh DD, Yin LX, Laaeq K, Merlo CA. A new endoscopic staging system for hereditary hemorrhagic telangiectasia. Int Forum Allergy Rhinol. 2014 Aug;4(8):635-9. doi: 10.1002/alr.21339. Epub 2014 Apr 29. PMID 24782401
- See also: Osler- Weber-Rendu Disease (Hereditary Hemorrhagic Telangiectasia). — http://emedicine.medscape.com/article/2048472-overviw#a5
- See also: Vitamin D: fact sheet for health professionals. — http://ods.od.nih.gov/factsheets/VitaminD-HealthProfessional/